CLINICAL TRIAL: NCT00033683
Title: A Randomised Trial Of Standard Anthracycline-Based Chemotherapy With Fluorouracil, Epirubicin And Cyclophosphamide (FEC) Or Epirubicin And CMF (Epi-CMF) Versus FEC Followed By Sequential Docetaxel As Adjuvant Treatment For Women With Early Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Resected Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069311; ICR-TACT; EU-20109
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2005-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Methotrexate; Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill any tumor cells remaining after surgery. It is not yet known which combination chemotherapy regimen is more effective in treating resected stage I or stage II breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens in treating women who have resected stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival of women with completely resected stage I or II breast cancer adjuvantly treated with fluorouracil, epirubicin, and cyclophosphamide (FEC) or epirubicin followed by cyclophosphamide, methotrexate, and fluorouracil (EPI-CMF) versus FEC followed by sequential docetaxel.
* Compare the acute toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, estrogen receptor status (positive vs negative), and nodal status. Within 8 weeks after definitive surgery, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are assigned to 1 of 2 standard adjuvant chemotherapy regimens.

  * Regimen A: Patients receive fluorouracil, epirubicin, and cyclophosphamide (FEC) IV on day 1. Treatment repeats every 3 weeks for 8 courses.
  * Regimen B: Patients receive epirubicin IV on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive cyclophosphamide orally on days 1-14 or IV on days 1 and 8 and methotrexate IV and fluorouracil IV on days 1 and 8 (CMF). Treatment with CMF repeats every 4 weeks for 4 courses.
* Arm II: Patients receive 4 courses of adjuvant chemotherapy with FEC as in arm I, regimen A. Patients then receive sequential docetaxel IV over 1 hour once every 3 weeks for 4 courses.

Beginning within 4 weeks after completion of adjuvant chemotherapy, patients who are not concurrently enrolled in the Standardization of Breast Radiotherapy (START) trial receive localized radiotherapy once daily, 5 days a week, for 3-5 weeks, according to local practice.

Beginning within 4 weeks after completion of adjuvant chemotherapy, patients who are estrogen receptor and/or progesterone receptor positive receive oral tamoxifen once daily for at least 5 years.

Quality of life is assessed at baseline, before course 5, at 3-4 weeks after course 8, and then at 9, 12, 18, and 24 months after initiation of adjuvant chemotherapy.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 3,340 patients (1,670 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed completely resected, invasive breast cancer for which adjuvant chemotherapy is indicated
* No clinical or radiological evidence of locoregional or metastatic disease
* No locally advanced tumors at diagnosis, indicated by any of the following:

  * Fixed tumors
  * Peau d'orange skin changes
  * Skin ulceration
  * Inflammatory changes (T4 or T3b, N2 disease)
* No male breast cancer
* No prior invasive breast cancer or bilateral breast cancer
* Prior ductal carcinoma in situ or lobular carcinoma in situ is allowed
* Must begin study chemotherapy within 8 weeks after definitive surgery
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age:

* Over 18

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* At least 2 years

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin normal
* AST no greater than 1.5 times normal
* Alkaline phosphatase no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 10 years except surgically cured nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious medical illness that would limit life expectancy
* No psychiatric condition that would preclude informed consent
* No active uncontrolled bacterial, viral, or fungal infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* See Disease Characteristics
* No prior cytotoxic chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy (e.g., tamoxifen) during study chemotherapy
* No concurrent hormone replacement therapy

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since any prior unlicensed drugs
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Jane Banerji, Study Chair — Institute of Cancer Research, United Kingdom
Locations (69):
- U.Z. Gasthuisberg, Leuven, Belgium
- United Kingdom (68):
  - North Devon District Hospital, Barnstaple, England
  - Royal United Hospital, Bath, England
  - Queen Elizabeth Hospital at University of Birmingham, Birmingham, England
  - City Hospital - Birmingham, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Pilgrim Hospital, Boston, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Royal Free and University College Medical School, Hampstead, London, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital, Hull, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's Hospital, London, England
  - St. Georges Hospital Medical School, London, England
  - Charing Cross Hospital, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Mount Vernon Hospital, Northwood, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Oldchurch Hospital, Romford, England
  - Salisbury District Hospital, Salisbury, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Royal South Hants Hospital, Southampton, England
  - North Staffs Royal Infirmary, Stoke-on-Trent, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay Devon, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - New Cross Hospital, Wolverhampton, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Bronglais General Hospital - Ceredigion and Mid Wales NHS trust, Aberystwyth, Wales
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Glan Clywd District General Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital, Swansea, Wales

REFERENCES:
- [Result] Hopwood P, Ellis P, Barrett-Lee P, et al.: Impact on quality of life (QL) during chemotherapy (CT) of FEC-T compared to FEC or E-CMF: results from the UK NCRI taxotere as adjuvant chemotherapy trial (TACT). [Abstract] J Clin Oncol 23 (Suppl 16): A-661, 43s, 2005.
- [Derived] Kilburn LS, Aresu M, Banerji J, Barrett-Lee P, Ellis P, Bliss JM. Can routine data be used to support cancer clinical trials? A historical baseline on which to build: retrospective linkage of data from the TACT (CRUK 01/001) breast cancer trial and the National Cancer Data Repository. Trials. 2017 Nov 23;18(1):561. doi: 10.1186/s13063-017-2308-6. PMID 29179731